CLINICAL TRIAL: NCT02360085
Title: Does Heart Rate Variablity (HRV) Predict Hypotension on Induction in Patients Undergoing Surgery for Cervical Myelopathy ?
Brief Title: Does Heart Rate Variablity (HRV) Predict Hypotension in Patients Undergoing Cervical Myelopathy Surgery ?
Status: Completed | Type: Observational
Sponsor: Lashmi Venkatraghavan (Other)
Responsible Party: Sponsor-Investigator, Lashmi Venkatraghavan, Director, Neuroanesthesia, Toronto Western Hospital, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Other Study IDs: 14-8164
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Heart Rate Variability
Keywords: Cervical Myelopathy; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cervical myelopathy is commonly associated with degenerative spinal disease. Dysfunction of the autonomic nervous system is also evident in many cases of cervical myelopathy. Autonomic dysfunction may result in haemodynamic instability and hypotension under anaesthesia. It is important to maintain adequate mean arterial pressure in order to perfuse the spinal cord and prevent cord ischemia. Heart rate variability, the physiological variations of the differences between heart beats, has been used to diagnose autonomic dysfunction. In patients with cervical myelopathy it may enable the anaesthetist to predict hypotension thereby allowing for early treatment and prevention of spinal cord ischemia.

DETAILED DESCRIPTION:
Protocol

1. Standard perioperative management Routine standard preparation of the patients will be carried out as per the investigators institutional standard for all patients undergoing cervical spine surgery. All routine physiological monitoring (ECG, invasive arterial blood pressure, SPO2, end tidal CO2, temperature and depth of anaesthesia monitoring) will be performed. The induction of anesthesia will be performed with propofol (2-5 mg/kg), fentanyl (3mcg/Kg) and rocuronium (0.6 mg/kg) for intubation of the patient's trachea once peripheral nerve stimulation shows no muscle twitches.
2. Study protocol Before general anesthesia, following a 10 minute stabilization period with the patient lying supine and breathing at a rate of 12 - 15 breaths per minute, a 5 minute ECG recording will be obtained. ECG data will be downloaded onto a study laptop for later analysis using LabChart Software to determine HRV values. Hemodynamic data and depth of anaesthesia will be collected from the preinduction period until skin incision at 1 minute intervals. The study will be complete after skin incision.

Data Collection and Management Data Collection The following data will be collected: patient demographics, surgical data including position technique, number of levels, duration, anaesthetic data including agents used, hemodynamic measurements from preinduction to surgical incision, Japanese Orthopaedic Association Score. The incidence of hypotension and the number of interventions required to keep mean arterial blood pressure above 70 mmHg will be recorded.

Significance of the study Identifying patients at risk for hypotension can be useful to prevent hypotension and to prepare to treat hypotension sooner so that the risk of spinal cord ischemia can be minimized.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients, aged 18 - 70 years with the history of cervical myelopathy, presenting for anterior or posterior cervical decompression and fusion.

Exclusion Criteria:

1. Patients with arrhythmias or absence of sinus rhythm
2. Diabetic patients
3. Degenerative neurological disease e.g. Parkinson's disease
4. Complete SCI
5. Inherited autonomic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cervical myelopathy presenting for cervical spine surgery at Toronto Western Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lashmi Venkatraghavan, MD, Principal Investigator — Department of Anesthesia, Toronto Western Hospital. University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervical Myelopathy Undergoing Spine Surgery: This is a prospective, single-center, observational study in adult (aged 18-70 years) patients undergoing elective anterior or posterior cervical decompression and fusion for cervical myelopathy in our institution during the period from Sept 2017 to June 2018.
Period: Overall Study
Arm/Group | Cervical Myelopathy Undergoing Spine Surgery
Started | 65
Completed | 49
Not Completed | 16

BASELINE CHARACTERISTICS:
Population: In total 65 patients were recruited for the study and 16 patients were excluded. 49 patients were included for final analysis.
Arm/Group | Cervical Myelopathy Undergoing Spine Surgery
Number analyzed (Participants) | 49
Age, Customized [Mean (Standard Deviation); unit: years]
  Female | 55 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 49 patients were included for final analysis.
  Participants
    Female | 14
    Male | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 49
Cervical myelopathy [Count of Participants; unit: Participants]
  mild | 37
  moderate to severe | 12

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Variability (HRV)
Description: Difference between total power (ms2) of patients in the hypotension group compared to stable group
Time Frame: 1 day
Population: All data are presented as Median [Interquartile range]
Measure: Median (Inter-Quartile Range); unit: ms2
Groups:
- Hypotension Group: HRV analysis in hypotension group
- No Hypotension Group: HRV analysis in stable group
Arm/Group | Hypotension Group | No Hypotension Group
Number analyzed (Participants) | 37 | 12
ms2 | 1439 [637.9 to 3130.5] | 2191 [1229.5 to 2613.0]

2. Primary Outcome: HRV Indices
Description: Differences in HRV indices between hypotension group and no hypotension group
Time Frame: 1 day
Population: All data are presented as Median [Interquartile range]. VLF- very low frequency, LF-low frequency, HF- high frequency.
Measure: Median (Inter-Quartile Range); unit: ms2
Groups:
- Hypotension Group; No Hypotension Group: VLF, LF and HF analysis
Arm/Group | Hypotension Group | No Hypotension Group
Number analyzed (Participants) | 37 | 12
ms2
  VLF | 684.8 [411.8 to 1399.5] | 705.8 [566.8 to 1649.0]
  LF | 290.2 [143.6 to 1208.0] | 406.5 [236.3 to 934.7]
  HF | 109.7 [64.8 to 430.8] | 350.4 [185.7 to 1634.5]

3. Primary Outcome: Mean Arterial Pressure
Description: Preoperative Analysis Mean Arterial Pressure between hypotension group and no hypotension group
Time Frame: one day
Population: All data are presented as Median [Interquartile range]
Measure: Median (Inter-Quartile Range); unit: mmHg
Groups:
- Hypotension Group: Mean Arterial Pressure analysis in hypotension group
- No Hypotension Group: Mean Arterial Pressure analysis in no hypotension
Arm/Group | Hypotension Group | No Hypotension Group
Number analyzed (Participants) | 37 | 12
mmHg | 96.0 [89.8 to 102.3] | 104.3 [93.2 to 111.4]

4. Primary Outcome: HRV Indices Analysis
Description: Low frequency (LF)/High frequency Ratio
Time Frame: One day
Population: Low Frequency to High Frequency ratio. All data are presented as Median [Interquartile range].
Measure: Median (Inter-Quartile Range); unit: Ratio
Groups:
- Hypotension Group; No Hypotension Group: Low Frequency to High Frequency ratio
Arm/Group | Hypotension Group | No Hypotension Group
Number analyzed (Participants) | 37 | 12
Ratio | 3.33 [1.93 to 4.95] | 1.22 [0.22 to 1.86]

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse event observed
Groups:
- All Patients: Heart Rate Variability in Patients with Cervical Myelopathy
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT02360085/Prot_SAP_000.pdf